CLINICAL TRIAL: NCT04225182
Title: Evaluation of the Effectiveness of a Muscular Strengthening Protocol With an Instrumented Orthosis for Gonarthrosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-PP-19
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2022-08

CONDITIONS: Gonarthrosis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with instrumented Orthosis (Experimental): patient will follow 8 weeks of muscular strengthening with the orthosis connected to the phone app associated
  Interventions: Device: with instrumented Orthosis
- without instrumented Orthosis (Active Comparator): patient will follow 8 weeks of traditional muscular strengthening without orthosis
  Interventions: Device: traditional rehabilitation protocol

INTERVENTIONS:
Device: traditional rehabilitation protocol — muscular strengthening protocol with traditional rehabilitation protocol without orthosis
  Arms: without instrumented Orthosis
Device: with instrumented Orthosis — 8 weeks of muscular strengthening with the orthosis connected to the phone app associated
  Arms: with instrumented Orthosis

SUMMARY:
The management of knee osteoarthritis via a physical activity protocol for rehabilitation has convincing results. However, the effectiveness of these protocols could be improved with a connected instrumented knee brace with an exercise protocol adapted for the patient which is supervise by an online physiotherapist to check the progression during home-based rehabilitation.

DETAILED DESCRIPTION:
The management of knee osteoarthritis via physical activity protocol for rehabilitation has convincing results. The aim of this study is to determine the improvement of the effectiveness of a home-based rehabilitation with and without instrumented knee brace for moderated gonarthrosis patients.

The study will focus during one years on 80 moderated gonarthrosis patients with a Kellgren and Lawrence (K&L) score between 2 and 3, aged between 50 and 80. Each patient will practice an 8 weeks progressive home exercise program with 3 session per weeks. The effectiveness of this protocol will be quantified with a gait analysis with kinematics, kinetics and electromyography, before and after the progressive home exercise protocol. The statistical analysis will focus on ANOVA and correlation between control group and instrumented knee brace group.

ELIGIBILITY:
Inclusion Criteria:

* Person who signed informative consent
* Affiliated with the social security
* Male and female aged between 50 and 80
* Walk without assistance
* Smartphone's use

Exclusion criteria:

* Person under protective measure
* Orthopedics issues
* Neurologic issues (MMSE Test < 24)
* Knee or hip prothesis
* Person with NSAIDs and analgesics treatment with an effective intake less than 48 hours before the evaluation
* Predominant patello-femoral arthritis
* Symptomatic hip OA
* Knee infection
* Knee injuries

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-06-02 (Actual)

PRIMARY OUTCOMES:
Change External Knee Moment Abduction (EKAM) during gait cycle from baseline at 8 weeks after rehabilitation | At the baseline (inclusion) and after 8 weeks of muscular strengthening
  Assessment of knee external knee moment abduction

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GUERIN, MD, Principal Investigator — Nice University Hospital
Locations (1):
- CHU de Nice, Nice, France